CLINICAL TRIAL: NCT02480647
Title: Randomized Clinical Trial the Use of Levonorgestrel-releasing Intrauterine System Versus Etonogestrel Implant in Pelvic Pain Control in Women With Endometriosis
Brief Title: Clinical Trial the Use of Levonorgestrel-releasing Intrauterine System Versus Etonogestrel Implant in Endometriosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Luis Bahamondes, Carvalho NM, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 44827415200005404
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Levonorgestrel; etonogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- levonorgestrel & etonogestrel (Experimental): Levonorgestrel releasing intrauterine system
  Other names:
  Mirena.
  Interventions: Drug: Levonorgestrel
- etonogestrel (Active Comparator): Etonogestrel implant:
  Other name: Implanon Releasing 20μg/day.
  Interventions: Drug: Etonogestrel

INTERVENTIONS:
Drug: Levonorgestrel — 20μg/day.
  Other Names: levonorgestrel releasing intrauterine system; Mirena
  Arms: levonorgestrel & etonogestrel
Drug: Etonogestrel — 20μg/day.
  Other Names: Implanon
  Arms: etonogestrel

SUMMARY:
Randomized clinical trial the use of levonorgestrel releasing intrauterine system.

Objectives: To evaluate and compare the efficacy of- levonorgestrel releasing intrauterine system l(LNG-IUS) in relation to the subdermal implant releasing etonogestrel (ENG) in the control of chronic pelvic pain and / or dysmenorrhea in women endometriosis.

DETAILED DESCRIPTION:
Randomized clinical trial the use of levonorgestrel releasing intrauterine system.

Objectives: To evaluate and compare the efficacy of- levonorgestrel releasing intrauterine system (LNG-IUS) in relation to the subdermal implant releasing etonogestrel (ENG) in the control of chronic pelvic pain and / or dysmenorrhea in women with endometriosis.

Methods: Will be assessed 103 women, aged 18-45 years, diagnosis of endometriosis confirmed by laparoscopy or laparotomy that presents chronic pelvic pain and / or dysmenorrhea. The study will be experimental, randomized , (5' women will be allocated to the LNG-IUS and 52 women will use the implant subdermal ENG). Women will be invited to participate in the study on the day and having the Family Planning Clinic with pelvic pain complaints and / or dysmenorrhea with a confirmed diagnosis of endometriosis in search of inserting a LNG-IUS. That day will be invited to be allocated by lottery (through a system of computer generated randomization; with opaque and sealed envelopes), the group that will use LNG-IUS or subdermal implant ENG. At the inclusion in the study will be held the insertion of the LNG-IUS or ENG implant and on this day the pain will be evaluated by visual analogue scale (VAS) of pain and applied the evaluation questionnaire of endometriosis. It will be a calendar to record delivered daily bleeding and EVA for daily assessment of pain. Women will return each 30 days (± 3 days) where the pain of registration will be evaluated by EVA and will be collected the bleeding and delivered a new calendar for the next 30 days. The end of the study It is expected to 180 days post-insertion of the LNG-IUS or the implant and, in the latter evaluation, will again be applied questionnaire. Cancer antigen 125 (CA-125), CD23 and endometrial biopsy will be evaluated at baseline and at last follow-up ( +/- 180 days).

Inclusion criteria:

* Women aged 18 to 45
* Absence of pregnancy
* Patients with chronic pelvic pain and / or dysmenorrhea with pain scores ≥ 4 on EVA pain and surgical and histopathological diagnosis of endometriosis in 14 last three months to two years, according to the current classification of the American Society for Reproductive Medicine and
* Accept participate and sign the consent form and clarified.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 45
* Absence of pregnancy
* Patients with chronic pelvic pain and / or dysmenorrhea with pain scores ≥ 4 on EVA pain and surgical and histopathological diagnosis of endometriosis in 14 last three months to two years, according to the current classification of the American Society for Reproductive Medicine and Enzian classification.
* Accept participate and sign the consent form and clarified

Exclusion criteria:

* Current wish to get pregnant
* I just want to use the LNG-IUS as treatment
* Contraindication to the use of LNG-IUS: Current pelvic inflammatory disease or appellant; infection of the lower genital tract; infected abortion during the last 3 months; purulent cervicitis; uterine or cervical malignancy; bleeding abnormal uterine undiagnosed; congenital uterine anomalies or acquired conditions associated with increased susceptibility to infections; acute liver disease or liver tumors; hypersensitivity to LNG.
* Contraindications to the use of ENG implants: pregnancy or suspected pregnancy;
* Active venous thromboembolic disorder; presence or history of liver disease serious as liver function values have not returned to normal; progestogen dependent tumors; abnormal bleeding undiagnosed; hypersensitivity to any component of implante.
* Abusive use of alcohol and / or other illicit drugs.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Pelvic pain. Pain intensity measure: Self reported pain intensity daily. each item scored 0-10. | 6 months
  Self reported pain intensity in the morning, afternoon, evening and winch activity over. Each item is scored 0-10. ( 0=no pain; 10= pain as bad as can be.

SECONDARY OUTCOMES:
Uterine bleeding | 6 months
  Self reported uterine bleeding in the morning, evening and which activity over. Each item is noted in menstrual calendar. ( 0=no bleeding; 1= spotting; 2- light and 3= intense, noted by the participant in menstrual calendar daily
Cancer antigen 125 | Baseline and after 180 days
  Ca 125 will be evaluated at baseline and at last follow-up ( +/- 180 days).

CONTACTS AND LOCATIONS:
Overall Officials: Nelsilene Tavares, MD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Nelsilene Mota Carvalho, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Walch K, Unfried G, Huber J, Kurz C, van Trotsenburg M, Pernicka E, Wenzl R. Implanon versus medroxyprogesterone acetate: effects on pain scores in patients with symptomatic endometriosis--a pilot study. Contraception. 2009 Jan;79(1):29-34. doi: 10.1016/j.contraception.2008.07.017. Epub 2008 Sep 25. PMID 19041438
- [Background] Yisa SB, Okenwa AA, Husemeyer RP. Treatment of pelvic endometriosis with etonogestrel subdermal implant (Implanon). J Fam Plann Reprod Health Care. 2005 Jan;31(1):67-70. doi: 10.1783/0000000052972799. PMID 15720856
- [Background] Zomer MT, Ribeiro R, Trippia CH, Cavalcanti TC, Hayashi RM, Kondo W. [Correlation between serum Ca-125 levels and surgical findings in women with symptoms evocative of endometriosis]. Rev Bras Ginecol Obstet. 2013 Jun;35(6):262-7. doi: 10.1590/s0100-72032013000600005. Portuguese. PMID 23929199
- [Background] Gerlinger C, Schumacher U, Faustmann T, Colligs A, Schmitz H, Seitz C. Defining a minimal clinically important difference for endometriosis-associated pelvic pain measured on a visual analog scale: analyses of two placebo-controlled, randomized trials. Health Qual Life Outcomes. 2010 Nov 24;8:138. doi: 10.1186/1477-7525-8-138. PMID 21106059
- [Derived] Carvalho N, Margatho D, Cursino K, Benetti-Pinto CL, Bahamondes L. Control of endometriosis-associated pain with etonogestrel-releasing contraceptive implant and 52-mg levonorgestrel-releasing intrauterine system: randomized clinical trial. Fertil Steril. 2018 Nov;110(6):1129-1136. doi: 10.1016/j.fertnstert.2018.07.003. PMID 30396557